CLINICAL TRIAL: NCT06154850
Title: Effects of Virtual Reality on Brain Hemodynamic Activity in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Kartal Dr. Lütfi Kirdar City Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ATADEK 2022-14/06
Record Dates: First submitted 2023-11-20; First posted 2023-12-04 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Rheumatoid Arthritis; Virtual Reality
MeSH Terms: conditions — Chronic Pain; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality (Experimental): Individuals will wear the headset for 10 minutes while playing NatureTrek application
  Interventions: Other: Immersive virtual reality
- Non-immersive Virtual Reality (Active Comparator): Individuals will watch a video including scenes from NatureTrek application for 10 minutes.
  Interventions: Other: Non-immersive virtual reality

INTERVENTIONS:
Other: Immersive virtual reality — Oculus Quest 2 will be used with NatureTrek application for 10 minutes.
  Arms: Immersive Virtual Reality
Other: Non-immersive virtual reality — Patients will watch a video including scenes from NatureTrek application on a screen.
  Arms: Non-immersive Virtual Reality

SUMMARY:
Virtual reality systems have been applied in recent years to reduce pain intensity and fear of movement in individuals with acute and chronic pain. The main mechanism of virtual reality methods in pain control is to provide the effect of distraction from pain. Virtual reality systems allow the individuals to feel themselves in a different environment and shift their attention to the game they are playing or the virtual world created rather than the pain they feel. This is thought to be the main mechanism of pain control. However, the cortical mechanism of the reduction in pain caused by virtual reality methods, especially in individuals with chronic pain, has not been fully elucidated.

It is predicted that the integration of virtual reality methods into treatment protocols will gradually increase by time, especially as a result of the reflection of technological developments in clinical practice. At this point, fNIRS, which enables the assessment of the functionality of brain areas during movement, has the potential to reveal the response of the effect provided by virtual reality technology in the prefrontal cortex.

The aims of our study were to examine brain hemodynamic activity during the experience of non-immersive and immersive virtual reality environments and the change in pain intensity after virtual reality applications in individuals with rheumatic diseases with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis,
* Right hand dominant,

Exclusion criteria:

* A history of acute pain up to 3 days prior to the date of evaluation,
* Any psychiatric and neurological diagnosis,
* Have a cognitive problem that prevents them from adapting to the working procedure,
* Using centrally acting medications and anti-depressants.
* Presence of neuropathic pain,
* Presence of vision or hearing problems,
* Any psychiatric and neurological diagnosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Functional near infrared spectrosopy | During the intervention
  Real-time measurement and monitoring of brain hemodynamics will be performed with a 24-channel fNIRS device (Brite 24, Artinis, The Netherlands). Recordings will be obtained with sensors placed in the prefrontal cortex. In the study design, after the sensors are placed on the scalp, a 1-minute recording will first be taken in the resting position. Afterwards, painful and painless mechanical stimuli will be given to the subjects during the viewing of fully immersive and non-immersive virtual reality environments.
Numeric Pain Rating Scale | Immediately after the intervention
  Numeric Pain Rating Scale will be used to quantify pain severity after both virtual reality applications. Patients will be asked to report their pain numerically as 0: no pain; 10: unbearable pain.

SECONDARY OUTCOMES:
Perceived Level of Fun | Immediately after the intervention
  The level of entertainment perceived by the participants after each virtual reality application will be evaluated on a scale of 0 to 10 (0 = not entertained at all, 10 = very entertained).
Heart rate variability | During the intervention
  Heart rate variability will be assessed using a wearable belt (Polar OH1 heart rate monitor).

OTHER OUTCOMES:
Pain Catastrophizing Scale | Pre-intervention
  Pain Catastrophizing Scale assesses catastrophic feelings associated with pain, is a Likert-type self-assessment scale consisting of 13 items rated between 0 and 4 points. The total score ranges from 0 to 52 and includes rumination, magnification and helplessness subscales. Higher scores on the scale indicate higher levels of pain catastrophizing.
Tampa Kinesiophobia Scale | Pre-intervention
  Tampa Kinesiophobia Scale consists of 17 questions and is used to assess fear and avoidance behaviors in diseases related to musculoskeletal injuries. The scale uses a 4-point Likert scoring system (1=strongly disagree and 4=strongly agree). The total score is calculated after reversing questions 4, 8, 12 and 16 and ranges from 17 to 68. Higher scores indicate higher levels of kinesiophobia.
Adverse effects | Immediately after the intervention
  VR related events included dizziness, nausea, eye strain, and seizure.
Pain Detect Questionnaire | Pre-intervention
  PainDETECT is a validated self-report tool to identify neuropathic pain features in a range of conditions. Pain Detect Questionnaire consists of 17 questions, and the maximum score is 30. Scores equal or above 19 indicate the presense of likely neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Mehmet Ali Aydınlar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No